CLINICAL TRIAL: NCT00097760
Title: Safety Study of Natalizumab in Combination With Glatiramer Acetate (GA)
Brief Title: Natalizumab in Combination With Glatiramer Acetate (GA) in Patients With Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-1803
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; MS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Natalizumab 300 mg, IV infusion, every 4 weeks in addition to 20 mg of glatiramer acetate SC, daily, for up to 20 weeks.
  Interventions: Drug: Natalizumab
- Group 2 (Placebo Comparator): Placebo, by IV infusion, every 4 weeks in addition to 20 mg glatiramer acetate, by SC injection, daily, for up to 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natalizumab — Natalizumab 300 mg, IV infusion, every 4 weeks in addition to 20 mg of glatiramer acetate SC, daily, for up to 20 weeks.
  Other Names: Tysabri
  Arms: Group 1
Drug: Natalizumab — Natalizumab, 300 mg IV infusion, every 4 weeks for up to 20 weeks.
  Other Names: Tysabri
  Arms: Group 1
Drug: Placebo — Placebo, by IV infusion, every 4 weeks in addition to 20 mg glatiramer acetate, by SC injection, daily, for up to 20 weeks.
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine if natalizumab in combination with Glatiramer Acetate (GA) is safe and effective in delaying progression of individuals diagnosed with relapsing-remitting Multiple Sclerosis (MS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS as defined by McDonald et al., criteria # 1-4
* Between the ages of 18 and 55, inclusive
* Baseline EDSS score between 0.0 and 5.0, inclusive
* Have been treated with GA for at least the 12 months prior to randomization

Exclusion Criteria:

* Primary progressive, secondary progressive or progressive relapsing MS
* MS relapse has occurred within the 50 days prior to randomization
* A clinically significant infectious illness
* History of, or abnormal lab result indicative of significant disease that would preclude the administration of a recombinant humanized antibody immunomodulating agent or GA for 20 weeks.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2003-06; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Rate of development of new active lesions on MRI scans. | Week 20

SECONDARY OUTCOMES:
Incidence and severity of adverse events. | Week 20

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, MD, Study Director — Biogen

REFERENCES:
- See also: The website of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families, and healthcare providers. — http://www.nationalmssociety.org
- See also: MSActiveSource.com is a resource for news, information, and disease management for all individuals touched by Multiple Sclerosis. This site is sponsored by Biogen. — http://www.msactivesource.com